CLINICAL TRIAL: NCT00045838
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA006-00-VP, In Uninfected Adult Volunteers
Brief Title: HIV-1 Vaccine Test in Uninfected Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study product was revised. PI withdrew the study without enrolling participants..
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020279; 02-I-0279
Record Dates: First submitted 2002-09-10; First posted 2002-09-11 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Healthy; HIV-Negative; Placebo Controlled; Volunteer; Dose-Escalation; Healthy Volunteers; HV; HIV Seronegativity; HIV Preventive Vaccine

INTERVENTIONS:
Drug: VCR-HIVDNA006-00-VP

SUMMARY:
This study will test the safety of an experimental vaccine against HIV and examine whether it induces an immune response to HIV. A vaccine is a substance given to try to create resistance or immunity to a disease or infection. The vaccine in this study is made from DNA (genetic material) of four HIV proteins called gag, pol, Nef, and Env. Injected into a human, the viral DNA instructs the body to make small amounts of some HIV proteins. This study will see if the body then creates an immune response to these proteins. Study participants cannot catch HIV or AIDS from the DNA vaccine or any proteins made from it.

Healthy normal volunteers between 18 and 60 years of age may be eligible for this study. Candidates will provide a medical history, including information on sexual behaviors and drug use. They will have a physical examination and blood and urine tests. Women will also have a pregnancy test. Women enrolled in the study must either be infertile (e.g., due to menopause or hysterectomy) or must agree either to abstain from heterosexual sex or to practice birth control for at least 21 days before beginning the study and throughout its duration.

Participants will be randomly assigned to receive either the experimental vaccine or a placebo (a control substance made up of an inactive salt solution) and will be divided into three groups, based on their entry into the study. Of the first seven people enrolled (Group 1), five will receive a 2-mg dose of vaccine and two will receive placebo. If the vaccine is safe at this dose, then in Group 2, five people will receive a 4-mg dose of vaccine and two will receive placebo. If this dose is safe, then in Group 3, thirty people will receive an 8-mg dose of vaccine and six will receive placebo.

All participants will receive three injections in an upper arm muscle-one injection a month for three months-with a needle-less device called a Biojector 2000® (Registered Trademark). At the time of each injection, participants will be observed for at least 1 hour after immunization. At home, they will record their temperature and any symptoms they may experience, including any effects at the injection site, for at least 2 days, or as long as the symptoms remain. If symptoms occur, participants will report them immediately to the clinic staff and, if necessary, come to the clinic for an examination.

Participants will have about 10 clinic visits during the study. Most visits will last about 2 hours; those on vaccination days will last about 4 hours. At each visit, participants will be checked for health changes or problems and will be asked about medications they are taking. Blood will be drawn for immune system testing. Additional laboratory tests may be requested between visits. Participants will be tested several times for HIV, will be questioned about their sexual behavior and drug use, and about social effects they may have experienced from their participation in the study.

Some of the blood drawn for this study will be used to test for HLA type-a genetic test of immune system markers. For research, HLA testing is sometimes used to try to identify factors associated with the progression of HIV disease or related conditions.

DETAILED DESCRIPTION:
This is a Phase I, randomized, controlled, double-blinded, dose-escalation study to examine tolerability, dose, and immune response of an HIV DNA plasmid vaccine. The hypothesis is that this vaccine will be safe for human administration and elicit immune responses to HIV. The primary objective is to evaluate the safety and tolerability in humans of VCR-HIVDNA006-00-VP and secondary objectives are to evaluate the immuogenicity of the vaccine and social impact of participating in an HIV-1 vaccine trial. A Data and Safety Monitoring Board (DSMB) will review protocol results twice prior to dose escalation to the 8 mg dose level.

ELIGIBILITY:
INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 60 years old.
2. Available for follow-up for the duration of the study (12 months).
3. Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
4. Able and willing to sign the informed consent form.
5. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
6. Willing to have blood samples used for future research.
7. Willing to complete questionnaire to identify HIV infection risks and amendable to risk reduction counseling.
8. In good general health without clinically significant medical history.
9. Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

   Laboratory Criteria within 28 days prior to enrollment:
10. Hematocrit greater than or equal to 34% for women; greater than or equal to 38% for men
11. WBC count: Non-African Americans equals 3,300-12,000 cells/mm(3); African-Americans equals 2,500-12,000 cells/mm(3) (in absence of clinical or pathological etiology)
12. Differential either within institutional normal range or accompanied by site physician approval
13. Total lymphocyte count: Non-African Americans greater than or equal to 800 cells/mm(3); African Americans greater than or equal to 650 cells/mm(3) (in the absence of clinical or pathological etiology)
14. Platelets equals 125,000-550,000/mm(3)
15. ALT (SGPT) less than or equal to 1.5 X upper limit of normal
16. Serum creatinine less than or equal to 1.4 mg/dL
17. Normal urinalysis defined as negative glucose, negative or trace protein, and negative or trace hemoglobin.
18. Negative FDA-approved HIV blood test
19. Negative Hepatitis B surface antigen
20. Negative anti-HCV or negative HCV PCR if the anti-HCV is positive

    Female-Specific Criteria:
21. Negative beta-HCG pregnancy test for women presumed to be of reproductive potential.
22. A female participant must meet one of the following criteria:

No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation.,

Or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and throughout the duration of the study,

Or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and throughout the duration of the study by one of the following methods:

condoms, male or female, with or without a spermicide

diaphragm or cervical cap with spermicide

intrauterine device

contraceptive pills, Norplant, or Depo-Provera

male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following is true.

Women:

1. Woman who is breast-feeding.

   Volunteer has received any of the following substances:
2. HIV vaccines in a prior clinical trial
3. Immunosuppressive or cytotoxic medications within the past six months with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteriods for an acute uncomplicated dermatitis
4. Blood products within 120 days prior to HIV screening
5. Immunoglobulin within 60 days prior to HIV screening
6. Live attenuated vaccines within 30 days prior to initial study vaccine administration
7. Investigational research agents within 30 days prior to initial study vaccine administration
8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration
9. Current anti-TB prophylaxis or therapy

   Volunteer has a history of any of the following clinically significant conditions:
10. Serious adverse reactions of vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
11. Autoimmune disease or immunodeficiency
12. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteriods.
13. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
14. Thyroid disease including history of thyroidectomy and diagnoses that required medication within the past 12 months.
15. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.
16. Hypertension that is not well controlled by medication or is more than 150/100 at enrollment.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Syphilis infection that is active or positive serology due to a syphilis infection treated less than six months ago.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study is eligible.
20. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring prolonged treatment more than 3 years ago.
21. Asplenia or any condition resulting in the absence or removal of the spleen.
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment.
23. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgement of the investigator, would interfere with or serve as a contraindication to protocol adherence or a volunteer's ability to give informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-08; Primary Completion 2003-04 (Estimated); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Stribling R, Brunette E, Liggitt D, Gaensler K, Debs R. Aerosol gene delivery in vivo. Proc Natl Acad Sci U S A. 1992 Dec 1;89(23):11277-81. doi: 10.1073/pnas.89.23.11277. PMID 1454808
- [Background] Tang DC, DeVit M, Johnston SA. Genetic immunization is a simple method for eliciting an immune response. Nature. 1992 Mar 12;356(6365):152-4. doi: 10.1038/356152a0. PMID 1545867
- [Background] Fynan EF, Webster RG, Fuller DH, Haynes JR, Santoro JC, Robinson HL. DNA vaccines: protective immunizations by parenteral, mucosal, and gene-gun inoculations. Proc Natl Acad Sci U S A. 1993 Dec 15;90(24):11478-82. doi: 10.1073/pnas.90.24.11478. PMID 8265577